CLINICAL TRIAL: NCT06781554
Title: Evaluation of the Performance and Safety of a Type I Collagen-Based Medical Device (MD-Small Joints Collagen Medical Device) i the Treatment of RHIZOARTROSIS. "SMAGENART PILOT STUDY"
Brief Title: Evaluation of the Performance and Safety of a Type I Collagen-Based Medical Device (MD-Small Joints Collagen Medical Device) i the Treatment of RHIZOARTROSIS
Acronym: SMAGENART
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guna S.p.a (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDG20232202
Record Dates: First submitted 2024-11-20; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-12

CONDITIONS: Trapeziometacarpal Osteoarthritis; Rhizarthrosis; MEDICAL DEVICE; Infiltrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MD-Small Joints Collagen Medical Device (Experimental): MD-Small Joints Collagen Medical Device intra/peri-articular infiltration of MD-Small Joints Collagen Medical Device will be performed The Investigation Plan envisages a single experimental group which will be treated with infiltrations of: MD-Small Joints Collagen Medical Device (GUNA, Milan-Italy).
  Composition per 2ml: collagen of porcine origin 100 µg Excipients: Violet, NaCl, Water for injection. The subjects will be treated with 1 infiltration with a volume of 2ml at the time of enrollment (T0) and on a weekly basis for a total of 5 infiltrations.
  Interventions: Device: MD-Small Joints Collagen Medical Device

INTERVENTIONS:
Device: MD-Small Joints Collagen Medical Device — The infiltrations will be performed using 2.5ml syringes and 26 gauge/13mm needles under complete aseptic conditions. The first 3 infiltrations will be carried out at both intra- and peri-articular levels by injecting MD-Small Joints Collagen Medical Device into the trapeziometacarpal joint until a counter-pressure is felt, preventing further penetration of the liquid; the remaining quantity (usually about 1ml) will be injected at the peri-articular level by retracting the needle tip. The fourth and fifth infiltrations will be performed only at the peri-articular level.

SUMMARY:
Collagen is a structural protein biopolymer consisting of three polypeptide chains wrapped around to form a right-handed triple helix. Its structure, characterized by the presence of glycine every third residue, a high content of proline and hydroxyproline, is stabilized by interchain hydrogen bonds and electrostatic interactions, giving the molecules high mechanical resistance, incompressibility, and simultaneously, extensibility, plasticity, and flexibility, making tissues abundant in collagen particularly resistant to stress and load. In humans, collagen is present especially in the skin, subcutaneous tissue, cartilage, bone, joint capsule, tendons, muscles, and ligaments.

Growing evidence supports the infiltrative use of type I collagen in the treatment of musculoskeletal pathologies. In particular, the intra-articular and peri-articular use of collagen has been proposed in the treatment of osteoarthritis in various body districts with the intention of limiting joint hypermobility, stabilizing the structure of joint and peri-articular components, reducing pain, and consequently improving function. Several clinical studies have demonstrated that its intra-articular infiltrative use could result in pain reduction and improvement of functionality in various cases of gonarthrosis and coxarthrosis. Regarding the conservative management of symptomatic thumb base osteoarthritis, some studies, albeit on limited case series, have highlighted how the use of type I collagen at the joint and peri-articular level can lead to better control of painful symptoms, improvement in functionality, and reduction of joint instability.

Recently, Randelli F. et al. studied the in vitro effects on tenocytes induced by type I swine collagen (MD-Tissue Collagen Medical Device). In vitro results seem to demonstrate that this medical device can induce proliferation and migration of tenocytes and synthesis, maturation, and secretion of type I collagen, favoring tendon repair.

Randelli F. et al. also demonstrated the mainly mechanical activity of MD-Tissue Collagen Medical Device, which is able to induce modifications of morpho-functional properties of tenocytes.

In this Clinical Investigation, we aim to investigate the performance and safety of an injectable medical device based on type I collagen of swine origin called MD-Small Joints Collagen Medical Device, in the treatment of symptomatic thumb base osteoarthritis.

The purpose of this research project is to understand through a multicenter Clinical Investigation, the performance and safety of an intra-articular and peri-articular treatment with a medical device (MD-Small Joints Collagen Medical Device) based on type I collagen in terms of pain reduction and joint function recovery in subjects with symptomatic thumb base osteoarthritis. The primary endpoint will consist of evaluating, through the Visual Analogue Scale (VAS), the performance of MD-Small Joints Collagen Medical Device in reducing pain associated with trapeziometacarpal osteoarthritis, at time T6 weeks (T6w) compared to T0 (day0). A reduction of at least 30% in the VAS score is considered clinically significant.

Secondary endpoints will consist of evaluating the performance of MD-Small Joints Collagen Medical Device through:

* VAS score assessment at T3 week and T16week /FU compared to T0;
* Disability of the Arm Shoulder and Hand score assessment at T6 week and T16 week /FU compared to T0 (day0);
* Functional Index for Hand Osteoarthritis assessment at T6 week and T16 week /FU compared to T0;
* Pinch Strength Test assessment at T6 week and T16 week/FU compared to T0;
* Evaluation of analgesic drug consumption through clinical diary in various study phases;
* Assessment of Adverse Event incidence.

DETAILED DESCRIPTION:
The purpose of this research project is to understand through a multicenter Clinical Investigation, the performance and safety of an intra-articular and peri-articular treatment with a medical device (MD-Small Joints Collagen Medical Device) based on type I collagen in terms of pain reduction and joint function recovery in subjects with symptomatic thumb base osteoarthritis.

STUDY DESIGN:

This multicenter pilot Clinical Investigation will be based on a One-sample design. Variables will be assessed at 4 different time points: baseline (T0), after 3 weeks (T3w), after 6 weeks (T6 weeks), and after 16 weeks (T16w/FU), which is 12 weeks after the end of the infiltrative treatment.

Subjects will be treated with one infiltration of 2ml volume at the time of enrollment (T0) and weekly for a total of 5 infiltrations.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged between 18 and 75 years;
* Subjects with clinically diagnosed symptomatic thumb carpometacarpal osteoarthritis confirmed radiographically (stages I and II according to Eaton and Littler's classification);
* [N.B. in case of bilateral symptomatic thumb carpometacarpal osteoarthritis, treatment can be unilateral only, at the level of the thumb carpometacarpal joint that is more affected at the time of enrollment].
* Subjects with a VAS score ≥ 5; [The request for pain intensity (VAS) from the patient should refer to moments of hand use, nota t rest!]
* Subjects with joint pain for at least 1 month;
* Subjects not using thumb carpometacarpal orthotic devices;
* Subjects agreeing not to take analgesics within 24 hours before the scheduled visits;
* Subjects capable of understanding and signing the Informed Consent.

Exclusion Criteria

* Subjects with rheumatological conditions involving the hands;
* Subjects who have undergone hand surgery for the affected pathology;
* Subjects who have received HA injections in the thumb carpometacarpal joint in the last 3 months;
* Subjects who have taken NSAIDs in the last 7 days and/or corticosteroids in the last 30 days;
* Subjects undergoing physical therapy such as X-ray therapy, Tecar therapy, shock wave therapy, laser therapy, ultrasound therapy in the last 3 months;
* Subjects with neoplastic pathology;
* Subjects with systemic infections;
* Subjects with uncontrolled diabetes;
* Subjects with neurological conditions that may affect active participation in the study;
* Subjects with coagulopathies or taking anticoagulants (vitamin K antagonists, heparin);
* Subjects undergoing immunosuppressive treatment;
* Subjects using drugs or abusing alcohol;
* Subjects allergic to porcine collagen;
* Female subjects who are pregnant or breastfeeding;
* Subjects participating in other clinical studies during the same period;
* Subjects unable to cooperate or for whom poor compliance is expected;
* Any condition that, in the investigator's judgment, recommends the subject's exclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2025-12-29 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
The performance of MD-Small Joints Collagen Medical Device in reducing pain | T6 week compared to T0 (day0)
  The primary endpoint will consist of evaluating, through the Visual Analogue Scale (VAS), the performance of MD-Small Joints Collagen Medical Device in reducing pain associated with trapeziometacarpal osteoarthritis at T6 weeks (T6w) compared to T0 (day0). A reduction in VAS score of at least 30% is considered clinically significant.

SECONDARY OUTCOMES:
evaluating the VAS performance of MD-Small Joints Collagen Medical Device | VAS at T3 week and T16week/FU compared to T0 (day 0);
  The secondary endpoints will include evaluating the VAS performance of MD-Small Joints Collagen Medical Device
Evaluating DASH performance of MD-Small Joints Collagen Medical Device | DASH at T6 week and T16week /FU compared to T0(day0);
  Evaluating DASH performance of MD-Small Joints Collagen Medical Device at T6 week and T16 week/FU compared to T0 (day0);
Evaluating FIHOA performance of MD-Small Joints Collagen Medical Device | FIHOA at T6 week and T16 week/FU compared to T0 (day0); .
  Assesments FIHOA at T6 week and T16week/FU compared to T0 (day0);
  .
Evaluation of Pinch Strength Test | Pinch Strength Test at T6 week and T16week /FU compared to T0 (day0);
  Pinch Strength Test at T6 week and T16week /FU compared to T0 (day0);
Consumption of analgesics during various stages of the study; | Baseline (T0), Week 1 (T1), Week 2 (T2), Week 3 (T3), Week 4 (T4) week 6 (T6) and week 16 (T16)
  Consumption of analgesics during various stages of the study;
Incidence of AE | Baseline (T0), Week 1 (T1), Week 2 (T2), Week 3 (T3), Week 4 (T4) week 6 (T6) and week 16 (T16)
  Incidence of Adverse Events

CONTACTS AND LOCATIONS:
Locations (1):
- ASST Grande Ospedale Metropolitano Niguarda Piazza dell'Ospedale Maggiore,, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2023-09-21): https://cdn.clinicaltrials.gov/large-docs/54/NCT06781554/Prot_000.pdf